CLINICAL TRIAL: NCT03825081
Title: Effectiveness of Pilocarpine and Brimonidine to Improve Near Visual Acuity in Patients With Monofocal Intraocular Lenses
Brief Title: Pilocarpine and Brimonidine in Patients With Monofocal Lenses
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-151H
Record Dates: First submitted 2019-01-21; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Presbyopia; Pseudophakia
MeSH Terms: conditions — Presbyopia; Pseudophakia | interventions — Brimonidine Tartrate; Pilocarpine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention (Experimental): Interventions will be the drugs:
  * pilocarpine - 0.5%
  * brimonidine - 0.2%
  One drop of each of the study drugs will be placed in the non-dominant eye and patient will be evaluated for adverse events. At hour 1 and 3 vision will be measured for distance at 20 ft and reading at 14 inches; pupil size will be measured and patient will be evaluated for adverse events. At hour 6 vision will be measured for distance at 20 ft and reading at 14 inches; pupil size will be measured; patient will be evaluated for adverse events; and quality of life/satisfaction survey (NEI RQL-42) will be given to patient.
  Interventions: Drug: Brimonidine, pilocarpine

INTERVENTIONS:
Drug: Brimonidine, pilocarpine — 1 drop of pilocarpine (0.5%)
  1 drop of brimonidine (0.2%)
  Other Names: Mirvaso; Alphagan P; Salagen; Isopto Carpine

SUMMARY:
The current study aims to assess the use of pilocarpine and brimonidine to improve near visual acuity in patietns with monofocal intraocular lenses. Thirty-three subjects with be enrolled and baseline visual acuity with be measured at near and distance. This will be compared to visual acuity after drop administration over 6 hours. A quality of life questionnaire will also be evaluated.

DETAILED DESCRIPTION:
This research study will try to find out if pilocarpine and brimonidine can help people with intraocular lens implants read without reading glasses. Thirty-three subjects will take part in this research study. Baseline visual acuity with be measured at near and distance. This will be compared to visual acuity after drop administration over 6 hours. A quality of life questionnaire will also be evaluated.All subjects will take part at Massachusetts Eye and Ear Infirmary (MEEI).

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet all of the inclusion criteria in order to be eligible to participate in the study. Men and women between ages 60 years and above with monofocal intraocular lenses bilaterally corrected for distance and +/- 0.5D sphere vision who need only +/- 2.5 D correction for reading. Given the age group selected only post menopausal women will be evaluated.

Exclusion Criteria:

* Individuals meeting any of the exclusion criteria at baseline will be excluded from study participation including: allergies to proparacaine, pilocarpine or brimonidine, eye infection or inflammation, glaucoma, retinal tear or retinal disease, eye surgery within the past 30 days, use of eye drops within the last seven days, participated in any other research study within the past 30 days. Patients using contact lenses.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in visual acuity after administration of pilocarpine and brimonidine | baseline; hour 1
  The primary aim of our study is to determine if the combination of pilocarpine and brimonidine improves near visual acuity in pseudophakic subjects 1 hour following drop placement, compared to baseline.

SECONDARY OUTCOMES:
Change in near and distance visual acuity | baseline; hours 1; 3; and 6
  Near visual acuity at 3 hours and 6 hours, distance visual acuity at 1,3, and 6 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gardiner, MD, Principal Investigator — Matthew_Gardiner@meei.harvard.edu
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No